CLINICAL TRIAL: NCT02965118
Title: Multi Center, Randomized, Double-blind, Placebo-controlled Parallel-group, Phase III Clinical Trial to Evaluate the Safety and Efficacy of PAC-14028 Cream in Mild to Moderate Atopic Dermatitis Patients
Brief Title: CAPTAIN-AD: Clinical Study of AmorePacific's TRPV1 Antagonist in Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amorepacific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAPTAIN-AD-301
Record Dates: First submitted 2016-11-14; First posted 2016-11-16 (Estimated); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PAC-14028 cream 1.0% (Experimental): PAC-14028 cream 1.0% will be applied to treatment area twice daily for 8 weeks.
  Interventions: Drug: PAC-14028 cream 1.0%
- PAC-14028 cream Vehicle (Placebo Comparator): PAC-14028 cream Vehicle will be applied to treatment area twice daily for 8 weeks.
  Interventions: Drug: PAC-14028 cream Vehicle

INTERVENTIONS:
Drug: PAC-14028 cream 1.0% — topical application
  Arms: PAC-14028 cream 1.0%
Drug: PAC-14028 cream Vehicle — topical application
  Arms: PAC-14028 cream Vehicle

SUMMARY:
This is a phase III study to investigate the safety and efficacy of PAC-14028 cream in Atopic Dermatitis patients.

DETAILED DESCRIPTION:
PAC-14028 cream 1.0% or placebo will be treated to Mild to Moderate Atopic Dermatitis patients twice daily for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 12 - 70 years.
* Who was diagnosed with Atopic Dermatitis according to Haniffin and Rajka criteria.
* Whose affected TBSA is over 5% and below 30%, and IGA score is 2 (mild) to 3 (moderate).
* Who voluntarily agreed to participate in the study and signed an informed consent form.

Exclusion Criteria:

* Who has skin diseases other than atopic dermatitis or scar in the affected area which can affect the study, determined by the study investigators.
* Who has clinically significant medical history or diseases involving liver, kidney, neurological system, psychical disorder that can affect study results.
* Who has used systemic steroids, antibiotics, immunosuppressants, or received phototherapy within 28 days before study drug administration.
* Who has used topical steroids, topical calcineurin inhibitors or antibiotics to treat atopic dermatitis within 14 days before study drug administration.
* Who has used or is expected to inevitably use prohibited concomitant medications during the study.
* Women who is pregnant /breast-feeding, or who has childbearing potential and does not use available contraceptives.
* Who has dosed other study medications within 30 days before screening.
* Who is determined ineligible for study participation by investigators for any other reasons.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2016-11; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Success rate of Investigator's Global Assessment (IGA) | 8 weeks
  Percent of patients with IGA score of 0 (clear) or 1 (almost clear)

SECONDARY OUTCOMES:
Change of Investigator's Global Assessment (IGA) score | 8 weeks
  Change of IGA score from baseline
Success rate of ≥2-grade Investigator's Global Assessment (IGA) | 8 weeks
  percent of patients with ≥2 grade reduction of IGA score
Percent of change in Eczema Area and Severity Index (EASI) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kyuhan Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No